CLINICAL TRIAL: NCT00257686
Title: Study Of Pitavastatin 1 Mg Vs. Pravastatin 10 Mg, Pitavastatin 2 Mg Vs. Pravastatin 20 Mg And Pitavastatin 4 Mg Vs. Pravastatin 40 Mg (Following Up-Titration) In Elderly Patients With Primary Hypercholesterolemia Or Combined Dyslipidemia
Brief Title: Study to Compare the Efficacy and Safety of Pitavastatin and Pravastatin in Elderly Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Europe (Industry)
Responsible Party: Neil Hounslow, Kowa Research Europe
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NK-104-306
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Hypercholesterolemia or Combined Dyslipidemia
Keywords: Kowa; Hypercholesterolemia; combined; dyslipidemia; elderly; pitavastatin; NK-104
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — pitavastatin; Pravastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Pitavastatin 1 mg (Experimental): Pitavastatin 1 mg once daily
  Interventions: Drug: Pitavastatin
- Pravastatin 10 mg (Active Comparator): Pravastatin 10 mg once daily
  Interventions: Drug: Pravastatin
- Pitavastatin 2 mg (Experimental): Pitavastatin 2 mg once daily
  Interventions: Drug: Pitavastatin
- Pravastatin 20 mg (Active Comparator): Pravastatin 20 mg once daily
  Interventions: Drug: Pravastatin
- Pitavastatin 4 mg (Experimental): Pitavastatin 4 mg once daily
  Interventions: Drug: Pitavastatin
- Pravastatin 40 mg (Active Comparator): Pravastatin 40 mg once daily
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pitavastatin
  Arms: Pitavastatin 1 mg; Pitavastatin 2 mg; Pitavastatin 4 mg
Drug: Pravastatin
  Arms: Pravastatin 10 mg; Pravastatin 20 mg; Pravastatin 40 mg

SUMMARY:
The purpose of this study is to compare the efficacy and safety of pitavastatin with that of pravastatin in elderly patients

DETAILED DESCRIPTION:
Following a wash-out dietary lead-in period, patients will receive either Preavastatin or Pitavastatin during 12 weeks, in order to establish the efficacy of pitavastatin in reducing cholesterol levels.

ELIGIBILITY:
Inclusion Criteria:

* Males and postmenopausal females (aged 65 years and older
* Eligible, able to participate, have given informed consent
* Must have been following a restrictive diet
* Diagnosis of primary hypercholesterolemia or combined dyslipidemia
* Serum CK must be less than or equal to 1.5 x ULRR at 2 of 3 permitted evaluations between Week -4 and -1
* Agree to be available

Exclusion Criteria

* Homozygous familial hypercholesterolemia
* Conditions which may cause secondary dyslipidemia
* Uncontrolled diabetes mellitus (HbA1c >8%).
* Any condition which might significantly alter the absorption, distribution, metabolism, or excretion of any drug.
* History of pancreatic injury or pancreatitis, or impaired pancreatic function/injury
* Liver injury
* Impaired renal function
* Current obstruction of the urinary tract or difficulty in voiding due to mechanical as well as inflammatory conditions, which is likely to require intervention during the course of the study or is regarded as clinically meaningful
* Serum CK >5 x ULRR without clinical explanation
* Uncontrolled hypothyroidism defined as TSH >ULRR
* Any severe acute illness or severe trauma in the last 3 months prior to Visit 1
* Major surgery, 3 months prior to Visit 1
* Significant CVD prior to randomization
* Evidence of symptomatic heart failure, gross cardiac enlargement; significant heart block or cardiac arrhythmias. History of uncontrolled complex ventricular arrhythmias, uncontrolled atrial fibrillation/flutter or uncontrolled supraventricular tachycardias with a ventricular response rate of > 100 beats per minute at rest.
* Left ventricular ejection fraction <0.25;
* History of symptomatic cerebrovascular disease
* Any other conditions at the discretion of the investigator
* Known HIV infection
* Poorly controlled or uncontrolled hypertension
* Prior or current known muscular or neuromuscular disease of any type;
* Neoplastic disease
* Drug abuse or continuous consumption of more than 65 mL pure alcohol per day
* Exposure to any investigational new drug within 30 days of study entry or ingestion of any drug known to be toxic to a major organ system
* Current or recent use of supplements known to alter lipid metabolism
* History of hypersensitivity to other HMG-CoA reductase inhibitors;
* Concomitant medication not permitted
* Resistant to lipid-lowering medications. Known hypersensitivity or intolerance to any lipid lowering agent
* Excessive obesity
* Any factor which makes regular clinic attendance in the morning impractical ---Signs of mental dysfunction or other factors likely to limit ability to cooperate with the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 962 (Actual)
Dates: Start 2005-09; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragos Budinski, MD, Study Director — Medical Director
Locations (62):
- Denmark (4):
  - CCBR A/S, Aalborg
  - Copenhagen University Hospital, Copenhagen
  - Medical Center, Copenhagen
  - CCBR A/S, Vejle
- Germany (18):
  - Kardiologische Gemeinschaftspraxis Prof. Reifart, Bad Soden / Taunus
  - Praxis Dr. Boenninghoff, Beckum
  - Klinische Forschung Berlin Mitte, Berlin
  - GWT-TUK mbH, Zentrum fur Klinische Studien, Dresden
  - Gemeinschaftspraxis Dr. Krause, Th. Menke, Goch
  - Klinische Forschung Hamburg, Hamburg
  - Innere Medizin I / Medizinische Klinik, Heidelberg
  - Gemeinschaftspraxis H. Holz Dr. med, K. W. Klingl, Lampertheim
  - ZET-Studien GmbH Leipzing, Leipzig
  - Internistische Gemeinschaftspraxis, Mainz
  - Praxis Dr. Wachter, Mannheim
  - Gemeinschaftspraxis Melcherstaette, Melcherstaette
  - Gemeinschaftspraxis Dr. Senftleber, Dr. Kohler, Messkirch
  - Praxisgemeinschaft im Kleinen Biergrund, Offenbach/M
  - Gemeinschaftspraxis Melcherstaette, Stuhr-Brinkum
  - Gemeinschaftspraxis Drs. Mockesch, Weinheim
  - Intermed Institud Fur Klinische Forschung und Arzn, Wiesbaden
  - Gemeinschaftspraxis Dr. Emden, Frank Drewes, Worpswede
- Israel (9):
  - Department of Internal Medicine, Soroka Medical Center, Beersheva
  - Department of Internal Medicine A, Rambal Medical Center, Haifa
  - Department of Internal Medicine, Wolfson Medical Center, Holon
  - Center for Research, Hadassah University Hospital, Jerusalem Ein Kerem
  - Meir Hospital, Kfar Saba
  - Department of Medicine, Hadassah Medical Center, Mount Scopus Jerusalem
  - Department of Internal Medicine, Rivka Sieff Medical Center, Safed
  - Institute of Metabolic Diseases, Tel Aviv
  - Institue of Lipid & Atherosclerosis Research, Tel Litwinsky
- Netherlands (11):
  - Andromed Oost, ES Velp
  - Andromed Noord, Groningen
  - Vasculair Onderzoek Centrum Hoorn, Hoorn
  - Andromed Leiden, Leiden
  - Andromed Nijmegen, Rotterdam
  - Andromed Rotterdam, Rotterdam
  - Albert Schweitzer ziekenhuis, Sliedrecht
  - Andromed Breda, VL Breda
  - Rivierenland Tiel, WP Tiel
  - Andromed Zoetermeer, Zoetermeer
  - Albert Schweitzer ziekenhuis, Zwijndrecht
- United Kingdom (20):
  - Oldfield Surgery, Bath
  - St James's Surgery, Bath
  - The Pulteney Practice, Bath
  - Birmingham Clinical Research Centre, Birmingham
  - Stonehill Medical Center, Bolton
  - Chorley Clinical Research Centre, Chorley
  - Saltash Health Center, Cornwall
  - Gomersal Lane Surgery, Dronfield
  - Townhead Research, Irvine
  - Crosby Clinical Research Centre, Liverpool
  - The Symons Medical Center, Maidenhead
  - Manchester Clinical Research Centre, Manchester
  - Greenwood Medical Center, Nottingham
  - Reading Clinical Research Centre, Reading
  - Elm Lane Surgery, Sheffield
  - Brook Lane Surgery, Southampton
  - Bradford Road Medical Center, Wiltshire
  - Rowden Medical Partnership, Wiltshire
  - The Porch Surgery, Wiltshire
  - The Burns Medical Practice, Yorkshire

REFERENCES:
- [Derived] Stender S, Budinski D, Gosho M, Hounslow N. Pitavastatin shows greater lipid-lowering efficacy over 12 weeks than pravastatin in elderly patients with primary hypercholesterolaemia or combined (mixed) dyslipidaemia. Eur J Prev Cardiol. 2013 Feb;20(1):40-53. doi: 10.1177/2047487312451251. Epub 2012 Jun 7. PMID 22679249

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pitavastatin 1 mg | Pravastatin 10 mg | Pitavastatin 2 mg | Pravastatin 20 mg | Pitavastatin 4 mg | Pravastatin 40 mg
Started | 209 | 108 | 226 | 99 | 216 | 104
Safety Population | 207 (Subjects who received at least one dose of study medication) | 103 (Subjects who received at least one dose of study medication) | 224 (Subjects who received at least one dose of study medication) | 96 (Subjects who received at least one dose of study medication) | 210 (Subjects who received at least one dose of study medication) | 102 (Subjects who received at least one dose of study medication)
Completed | 188 | 89 | 208 | 88 | 194 | 95
Not Completed | 21 | 19 | 18 | 11 | 22 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin 1 mg | Pravastatin 10 mg | Pitavastatin 2 mg | Pravastatin 20 mg | Pitavastatin 4 mg | Pravastatin 40 mg | Total
Number analyzed (Participants) | 207 | 103 | 224 | 96 | 210 | 102 | 942
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 207 | 103 | 224 | 96 | 210 | 102 | 942
Age Continuous [Mean (Standard Deviation); unit: years] | 70.0 (4.60) | 70.5 (4.61) | 70.5 (4.49) | 69.9 (4.51) | 70.2 (4.10) | 70.2 (4.94) | 70.2 (4.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 54 | 124 | 48 | 121 | 42 | 507
  Male | 89 | 49 | 100 | 48 | 89 | 60 | 435

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C
Description: Percent change from baseline in low density cholesterol (LDL-C)
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Pitavastatin 1 mg | Pravastatin 10 mg | Pitavastatin 2 mg | Pravastatin 20 mg | Pitavastatin 4 mg | Pravastatin 40 mg
Number analyzed (Participants) | 207 | 103 | 224 | 96 | 210 | 102
Percent change | -31.43 (11.833) | -22.41 (14.051) | -38.99 (13.069) | -28.83 (11.054) | -44.31 (13.695) | -33.98 (14.299)

2. Secondary Outcome: Percent Change From Baseline in TC
Description: Percent change from baseline in total cholesterol (TC)
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Pitavastatin 1 mg | Pravastatin 10 mg | Pitavastatin 2 mg | Pravastatin 20 mg | Pitavastatin 4 mg | Pravastatin 40 mg
Number analyzed (Participants) | 207 | 103 | 224 | 96 | 210 | 102
Percent change | -22.19 (8.899) | -15.34 (11.037) | -26.68 (9.429) | -20.61 (8.426) | -30.75 (10.461) | -24.07 (10.907)

ADVERSE EVENTS:
Arm/Group | Pitavastatin 1 mg | Pravastatin 10 mg | Pitavastatin 2 mg | Pravastatin 20 mg | Pitavastatin 4 mg | Pravastatin 40 mg
Serious Adverse Events (participants affected / at risk) | 1 | 0 | 2 | 1 | 3 | 3
Other Adverse Events (participants affected / at risk) | 59 | 36 | 62 | 24 | 52 | 23
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Pitavastatin 1 mg | Pravastatin 10 mg | Pitavastatin 2 mg | Pravastatin 20 mg | Pitavastatin 4 mg | Pravastatin 40 mg
Acute myocardial infarction (Cardiac disorders) | 0/207 | 0/103 | 0/224 | 0/96 | 0/210 | 1/102
Myocardial infarction (Cardiac disorders) | 0/207 | 0/103 | 0/224 | 0/96 | 1/210 | 0/102
Cholecystitis (Hepatobiliary disorders) | 0/207 | 0/103 | 0/224 | 0/96 | 0/210 | 1/102
Cholelithiasis (Hepatobiliary disorders) | 0/207 | 0/103 | 0/224 | 0/96 | 0/210 | 1/102
Concussion (Injury, poisoning and procedural complications) | 0/207 | 0/103 | 1/224 | 0/96 | 0/210 | 0/102
Femoral neck fracture (Injury, poisoning and procedural complications) | 0/207 | 0/103 | 0/224 | 0/96 | 1/210 | 0/102
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0/207 | 0/103 | 0/224 | 0/96 | 1/210 | 0/102
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0/207 | 0/103 | 0/224 | 0/96 | 1/210 | 0/102
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/207 | 0/103 | 0/224 | 1/96 | 0/210 | 0/102
Cerebral thrombosis (Nervous system disorders) | 1/207 | 0/103 | 0/224 | 0/96 | 0/210 | 0/102
Urinary incontinence (Renal and urinary disorders) | 0/207 | 0/103 | 1/224 | 0/96 | 0/210 | 0/102
Bleeding varicose vein (Vascular disorders) | 0/207 | 0/103 | 0/224 | 0/96 | 0/210 | 1/102
Hypertensive crisis (Vascular disorders) | 0/207 | 0/103 | 0/224 | 0/96 | 0/210 | 1/102
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pitavastatin 1 mg | Pravastatin 10 mg | Pitavastatin 2 mg | Pravastatin 20 mg | Pitavastatin 4 mg | Pravastatin 40 mg
Nasopharyngitis (Infections and infestations) | 15/207 | 6/103 | 16/224 | 5/96 | 19/210 | 7/102
Influenza (Infections and infestations) | 7/207 | 6/103 | 16/224 | 6/96 | 19/210 | 7/102
Upper respiratory infection (Infections and infestations) | 3/207 | 4/103 | 2/224 | 1/96 | 3/210 | 3/102
Constipation (Gastrointestinal disorders) | 10/207 | 5/103 | 6/224 | 4/96 | 9/210 | 3/102
Nausea (Gastrointestinal disorders) | 5/207 | 5/103 | 6/224 | 1/96 | 3/210 | 0/102
Myalgia (Musculoskeletal and connective tissue disorders) | 3/207 | 3/103 | 11/224 | 2/96 | 4/210 | 2/102
Back pain (Musculoskeletal and connective tissue disorders) | 6/207 | 3/103 | 9/224 | 1/96 | 3/210 | 2/102
Headache (Nervous system disorders) | 8/207 | 3/103 | 9/224 | 4/96 | 4/210 | 2/102
Fatigue (General disorders) | 2/207 | 4/103 | 0/224 | 0/96 | 4/210 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days